CLINICAL TRIAL: NCT00523653
Title: The Genetics of Dilated Cardiomyopathy: A Quebec-Based Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Dr Nadia Giannetti, McGill University Health Center
Other Study IDs: BMB 07-004
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Dilated Cardiomyopathy (DCM)
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood test — looking at DNA

SUMMARY:
Dilated cardiomyopathy (DCM) affects about 200,000 Canadians. Eighty percent of these cases are of unclear cause, often occuring in families. We believe that mutations in specific already-identified genes contribute to DCM in Quebec and that certain mutations may account for a significant proportion of cases due to the well-documented "founder effect". Two hundred patients with DCM followed in our Heart Function Clinic will be approached for one blood sample at their routine clinic visit to test this hypothesis. The samples will be tested in the Laboratory of Cardiovascular Genetics at the Royal Victoria Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Followed at MUHC Heart Function Centre
* Documented EF of less than or equal to 35% and an enlarged heart with a left ventricular end-diastolic size of greater than 6 cm.
* Patient's written consent

Exclusion Criteria:

* Patients with a known underlying condition that results in a weakened and enlarged heart
* Patients unable to read and understand the consent form
* Patients who do not wish to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Dilated cardiomyopathy followed at the Heart Function Clinic and their families
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia S Giannetti, MD, Principal Investigator — McGill University Hospital Centre; Jamie Engert, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada